CLINICAL TRIAL: NCT01031407
Title: Cognitive Neuroscience of Autism Spectrum Disorders
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 100027; 10-M-0027
Record Dates: First submitted 2009-12-11; First posted 2009-12-14 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2025-11-26

CONDITIONS: Asperger's Disorder; Mental Retardation; Children; Adult; Autism Spectrum Disorders
Keywords: Social Cognition; Autism; Functional Magnetic Resonance Imaging (fMRI); MEG; Structural MRI; Natural History
MeSH Terms: conditions — Asperger Syndrome; Intellectual Disability; Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Healthy Volunteers
- Group 2: Individuals with Autism Spectrum Disorders
- Group 3: Parents of Healthy Volunteers, or Individuals with Autism Spectrum Disorders

SUMMARY:
Background:

* Autism spectrum disorders (ASDs) are a group of developmental disorders that affect communication, social interaction, and behavior. Relatively little is known about the relationship between genetics and behavior among these individuals and their close relatives. Researchers are interested in using interviews and rating scales to better understand these issues, as well as collecting brain scan data and genetic samples for testing and comparison.
* By comparing test results and genetic samples from healthy volunteers, people with ASD, and parents (or caregivers or legal guardians) of the first two groups, researchers hope to better understand the neuroscience of ASD.

Objectives:

* To learn more about the brain in healthy people and in people with autism spectrum disorders.
* To study genes that might be involved in autism spectrum disorders by collecting DNA samples from participants.

Eligibility:

The following groups of participants will be eligible for the study:

* Individuals between 5 and 89 years of age who have autism spectrum disorders.
* Healthy volunteers between 5 and 89 years of age.
* Cognitively impaired children between 5 and 17 years of age.
* Parents/caregivers/legal guardians of individuals in the above three groups.

Design:

* Participants will visit the National Institutes of Health Clinical Center for research tests, which will be administered over multiple visits. Researchers will determine the specific tests to be administered based on the medical history of the study participant.
* Researchers will study the brain through interviews, tests of thinking and memory (neuropsychological tests), brain imaging with magnetic resonance imaging (MRI), and magnetoencephalography (MEG).
* The study will also collect blood or saliva to obtain a DNA sample.

DETAILED DESCRIPTION:
Objective: The primary objective of the proposed studies is to utilize neuroimaging (functional Magnetic Resonance Imaging [fMRI], structural MRI [sMRI], Magnetoencephalography [MEG]) and neuropsychological tools (eye-tracking, cognitive experiments, clinical neuropsychological measures, questionnaires, etc.) to identify cognitive idiosyncrasies (e.g., social-cognitive deficits, visual perceptual assets, and savant skills) characteristic of individuals on the autism spectrum and their neural underpinnings across childhood and adulthood.

Study Population: Children, adolescents, and adults with autism spectrum disorders (ASDs), controls (i.e., typically developing children, adolescents, and adults and those with mild to moderate mental retardation), as well as caregivers/legal guardians/parents of these individuals.

Design: Descriptive/Characterization/Observational studies using primarily neuropsychological and neuroimaging methodologies.

Outcome Measures: Behavioral (reaction time, accuracy, eye movements, etc.) and neuroimaging (brain morphometry, BOLD, electrophysiology, etc.).

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects will include:

1. males and females.
2. 5-89 years of age.
3. A minimum IQ of 70

Subjects in the ASD group will:

1. meet DSM-IV criteria for one of the pervasive developmental disorders (i.e., autistic disorder, Asperger disorder, or pervasive developmental disorder-not otherwise specified).
2. meet or pass the autism cut-off score for social symptoms on the ADI and/or the ASD cut-off score from social+communication symptoms on the ADOS.
3. be able to provide their own consent (for adults).

For inclusion in the facial recognition substudy, subjects must be:

1. ages 18 to 35
2. in good health
3. with bad memory of faces

EXCLUSION CRITERIA:

All subjects, except for savants, also will be excluded if they have:

1. a history of neurological insult/injury.
2. substantial prenatal drug exposure known to affect later brain and behavior (e.g., cocaine, alcohol).
3. severely premature birth or birth trauma.
4. severe medical disorder (e.g., neurofibromatosis, hydrocephalus, cerebral palsy, uncontrollable seizure disorder).
5. a known genetic disorder (e.g., Fragile X or Down syndrome) that would be expected to significantly impact findings from cognitive testing and/or neuroimaging.

   Furthermore, subjects will be excluded from MRI/MEG studies, if they have:
6. any exclusion from MRI scanning including: the presence of metal in their body, having a pacemaker, and/or females who are pregnant.

Healthy volunteers, except for parents of individuals with autism spectrum disorders and parents of healthy volunteers, will also be excluded if they have:

1. a current or past history of axis I psychiatric conditions or any current usage of psychiatric medication.

Savants have less restrictive exclusionary criteria because: 1) they are a very rare group, thus we don t want to limit recruitment further and 2) we can examine common and unique cognitive mechanisms across savants, a question of keen interest, regardless of co-morbidities. Those with tumors or other neuroimaging-relevant contraindications will be excluded from fMRI/MEG procedures.

Ages: 5 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children, adolescents, and adults with autism spectrum disorders (ASDs), controls (i.e., typically developing children, adolescents, and adults and children with mild to moderate intellectual disability), as well as caregivers/legal guardians/parents of these individuals.
Sampling Method: Non-Probability Sample
Enrollment: 678 (Actual)
Dates: Start 2010-02-21 (Actual)

PRIMARY OUTCOMES:
Cognitive and neurological phenotypes in ASD and control participants | Ongoing
  Cognitive tasks and neuroimaging

CONTACTS AND LOCATIONS:
Overall Officials: Christopher I Baker, Ph.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Lynch CJ, Silver BM, Dubin MJ, Martin A, Voss HU, Jones RM, Power JD. Prevalent and sex-biased breathing patterns modify functional connectivity MRI in young adults. Nat Commun. 2020 Oct 20;11(1):5290. doi: 10.1038/s41467-020-18974-9. PMID 33082311
- [Derived] Avery JA, Liu AG, Ingeholm JE, Riddell CD, Gotts SJ, Martin A. Taste Quality Representation in the Human Brain. J Neurosci. 2020 Jan 29;40(5):1042-1052. doi: 10.1523/JNEUROSCI.1751-19.2019. Epub 2019 Dec 13. PMID 31836661
- [Derived] Power JD, Lynch CJ, Gilmore AW, Gotts SJ, Martin A. Reply to Spreng et al.: Multiecho fMRI denoising does not remove global motion-associated respiratory signals. Proc Natl Acad Sci U S A. 2019 Sep 24;116(39):19243-19244. doi: 10.1073/pnas.1909852116. Epub 2019 Aug 27. No abstract available. PMID 31455743
- [Derived] Ramot M, Walsh C, Martin A. Multifaceted Integration: Memory for Faces Is Subserved by Widespread Connections between Visual, Memory, Auditory, and Social Networks. J Neurosci. 2019 Jun 19;39(25):4976-4985. doi: 10.1523/JNEUROSCI.0217-19.2019. Epub 2019 Apr 29. PMID 31036762
- [Derived] Smith REW, Avery JA, Wallace GL, Kenworthy L, Gotts SJ, Martin A. Sex Differences in Resting-State Functional Connectivity of the Cerebellum in Autism Spectrum Disorder. Front Hum Neurosci. 2019 Apr 5;13:104. doi: 10.3389/fnhum.2019.00104. eCollection 2019. PMID 31024276
- [Derived] Jasmin K, Gotts SJ, Xu Y, Liu S, Riddell CD, Ingeholm JE, Kenworthy L, Wallace GL, Braun AR, Martin A. Overt social interaction and resting state in young adult males with autism: core and contextual neural features. Brain. 2019 Mar 1;142(3):808-822. doi: 10.1093/brain/awz003. PMID 30698656
- [Derived] Crutcher J, Martin A, Wallace GL. Dissociations in the neural substrates of language and social functioning in autism spectrum disorder. Autism Res. 2018 Aug;11(8):1175-1186. doi: 10.1002/aur.1969. PMID 30365251
- [Derived] Avery JA, Ingeholm JE, Wohltjen S, Collins M, Riddell CD, Gotts SJ, Kenworthy L, Wallace GL, Simmons WK, Martin A. Neural correlates of taste reactivity in autism spectrum disorder. Neuroimage Clin. 2018 Apr 4;19:38-46. doi: 10.1016/j.nicl.2018.04.008. eCollection 2018. PMID 30035000
- [Derived] Power JD, Plitt M, Gotts SJ, Kundu P, Voon V, Bandettini PA, Martin A. Ridding fMRI data of motion-related influences: Removal of signals with distinct spatial and physical bases in multiecho data. Proc Natl Acad Sci U S A. 2018 Feb 27;115(9):E2105-E2114. doi: 10.1073/pnas.1720985115. Epub 2018 Feb 12. PMID 29440410
- [Derived] Power JD, Plitt M, Laumann TO, Martin A. Sources and implications of whole-brain fMRI signals in humans. Neuroimage. 2017 Feb 1;146:609-625. doi: 10.1016/j.neuroimage.2016.09.038. Epub 2016 Oct 15. PMID 27751941
- [Derived] Power JD. A simple but useful way to assess fMRI scan qualities. Neuroimage. 2017 Jul 1;154:150-158. doi: 10.1016/j.neuroimage.2016.08.009. Epub 2016 Aug 7. PMID 27510328
- [Derived] Eisenberg IW, Wallace GL, Kenworthy L, Gotts SJ, Martin A. Insistence on sameness relates to increased covariance of gray matter structure in autism spectrum disorder. Mol Autism. 2015 Oct 1;6:54. doi: 10.1186/s13229-015-0047-7. eCollection 2015. PMID 26435832
- [Derived] Martin A. GRAPES-Grounding representations in action, perception, and emotion systems: How object properties and categories are represented in the human brain. Psychon Bull Rev. 2016 Aug;23(4):979-90. doi: 10.3758/s13423-015-0842-3. PMID 25968087
- [Derived] Plitt M, Barnes KA, Martin A. Functional connectivity classification of autism identifies highly predictive brain features but falls short of biomarker standards. Neuroimage Clin. 2014 Dec 24;7:359-66. doi: 10.1016/j.nicl.2014.12.013. eCollection 2015. PMID 25685703
- [Derived] Kenworthy L, Wallace GL, Birn R, Milleville SC, Case LK, Bandettini PA, Martin A. Aberrant neural mediation of verbal fluency in autism spectrum disorders. Brain Cogn. 2013 Nov;83(2):218-26. doi: 10.1016/j.bandc.2013.08.003. Epub 2013 Sep 18. PMID 24056237
- [Derived] Gotts SJ, Jo HJ, Wallace GL, Saad ZS, Cox RW, Martin A. Two distinct forms of functional lateralization in the human brain. Proc Natl Acad Sci U S A. 2013 Sep 3;110(36):E3435-44. doi: 10.1073/pnas.1302581110. Epub 2013 Aug 19. PMID 23959883
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2010-M-0027.html